CLINICAL TRIAL: NCT00992797
Title: A Randomized Controlled Trial of the Effect of Vitamin D Supplementation on Insulin Sensitivity and Secretion in Subjects With Type 2 Diabetes of Nordic and Sub-Indian Ethnicity .
Brief Title: Diabetes Intervention Trial With Vitamin D in Subjects of Nordic and Sub-Indian Ethnicity
Acronym: DIVINE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Aker (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Director of Research Tomm Bernklev, Oslo University Hospital, Aker
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUS-KIB-001
Record Dates: First submitted 2009-10-05; First posted 2009-10-09 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-11

CONDITIONS: Diabetes Mellitus Type 2; Hypovitaminosis D
Keywords: Insulin resistance; Insulin secretory dysfunction; Inflammation; Vascular stiffness
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Vitamin D Deficiency; Insulin Resistance; Inflammation | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholecalciferol (Experimental)
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator)
  Interventions: Other: Orange juice

INTERVENTIONS:
Drug: Cholecalciferol — Cholecalciferol 200.000 IU pr ampoule, 400.000 IU given at randomization day, followed by additionally 200.000 IU at week 5 if serum 25(OH)D < 100 nmol/L. If serum 25(OH)D > 100 placebo will be given. The cholecalciferol will be given in orange juice.
  Other Names: Vitamin D; ZymaD
  Arms: Cholecalciferol
Other: Orange juice — Orange juice at randomization day and at week 5.
  Arms: Placebo

SUMMARY:
The aim of this 6 months study is to evaluate the metabolic effects of 400.000-600.000 IU of vitamin D supplementation in subjects with type 2 diabetes and hypovitaminosis D. The main hypothesis is that subjects with low levels of 25-OH-vitamin D will benefit from supplementation with cholecalciferol in sufficient doses to optimize serum levels.

DETAILED DESCRIPTION:
Accumulating evidence suggests that hypovitaminosis D may be associated with the development of type 2 diabetes and disturbances in glucose and insulin metabolism. There is lack of data from randomized, controlled studies of sufficient duration and with the use of sufficient doses of vitamin D to assess the importance of vitamin D supplementation in glucose metabolism in type 2 diabetes.

ELIGIBILITY:
Inclusion criteria:

1. Moderate (S-25OHD 25-50 nmol/l) to severe (S-25OHD < 25 nmol/l) vitamin D deficiency measured at Visit 1.
2. Patients with type 2 diabetes, including drug naïve subjects, subjects using oral anti-diabetic medication and subjects on insulin treatment. All medication must be in stable doses during the 4 week lead-in period.
3. HbA1c < 11 % at Visit 1.
4. Able to communicate in Norwegian.
5. Men and women ≥ 18 years.
6. Norwegian or South Asian ethnicity.
7. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study. All WOCBP must have negative serum or urine pregnancy test at enrollment, randomization, titration visit and final study assessment.
8. Antihypertensive medication, lipid lowering drugs, oral contraceptives, hormone replacement therapy, multivitamin supplements and nutritional supplements are allowed if the subjects adhere to the same regimen during the study

Exclusion Criteria:

1. Subjects not having type 2 diabetes.
2. SBP ≥ 160 or DBP ≥ 95 at Visit 1.
3. Significant renal disease or chronic renal impairment, GFR< 30 ml/min.
4. Significant liver disease or ASAT or ALAT >3x UNL.
5. Malignancy during the last five years.
6. Hypercalcemia at Visit 1.
7. A history of kidney stone disease
8. WOCBP unwilling or unable to use an acceptable method to avoid pregnancy.
9. Pregnant or breastfeeding women.
10. Chronic inflammatory disease in active phase
11. Long term (>2 weeks) use of corticosteroids last 3 months
12. Mental condition (psychiatric or organic cerebral disease) rendering the subject unable to understand the nature, scope and possible consequences of the study.
13. Drug or alcohol abuse.
14. BMI > 45 kg/m2 or bariatric surgery (<5 years).
15. Anemia
16. Cardiovascular disease (myocardial infarction, unstable angina pectoris or stroke) during the last 6 months.
17. Any medical condition that in the judgment of the investigator would jeopardize the subject's safety or evaluation of the study drug for efficacy and safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity measured with euglycemic, hyperinsulinemic clamp | Before and after the 6 months intervention period

SECONDARY OUTCOMES:
Insulin secretion measured with IVGTT | At 0 and 6 months
Physical activity/muscle strength | At 0 and 6 months
HbA1c and fasting glucose | At 0, 3 and 6 months
Arterial stiffness | At 0 and 6 months
Differences in inflammatory markers, endothelial function and bone specific laboratory markers. | At 0, 3 and 6 months
Safety of this regimen of vitamin D3 supplementation; subjects will be assessed for hypercalcemia and renal dysfunction. | Entire intervention period, samples taken at 0,1,3, and 6 months
Change from baseline in quality of life score between groups (SF-36). | At 0 and 6 months
Effect on serum lipid levels and other biochemical markers | At 0, 3 and 6 months
Metabolomics analyses. | At 0 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kåre I Birkeland, MD PhD, Principal Investigator — Oslo University Hospital, Aker
Locations (1):
- Diabetes Laboratory, Oslo University Hospital Aker, Oslo, Norway

REFERENCES:
- [Derived] Gulseth HL, Wium C, Angel K, Eriksen EF, Birkeland KI. Effects of Vitamin D Supplementation on Insulin Sensitivity and Insulin Secretion in Subjects With Type 2 Diabetes and Vitamin D Deficiency: A Randomized Controlled Trial. Diabetes Care. 2017 Jul;40(7):872-878. doi: 10.2337/dc16-2302. Epub 2017 May 3. PMID 28468770